CLINICAL TRIAL: NCT00515593
Title: Non-interventional Open Single Arm, Multicentre Study to Observe the Use of Preotact in Patients With Severe Postmenopausal Osteoporosis
Brief Title: PROPOSE Quality - PReOtact in Postmenopausal OStEoporosis - Quality of Life Study (FP-004-DE)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Other Study IDs: FP-004-DE
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Postmenopause; Osteoporosis
Keywords: osteoporosis; postmenopausal women; Severe postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Parathyroid Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Parathyroid hormone (PTH) (Preotact) — Patients with severe postmenopausal osteoporosis

SUMMARY:
The objectives of the study are

* to describe the quality of life at the beginning of the Preotact® treatment and at the end of the observational period (Qualeffo-41 questionnaire)
* pain assessment at the beginning of the Preotact® treatment and at the end of the observational period (VAS score)
* to describe bone mineral density at the beginning of the Preotact® treatment and at the end of the observational period (T-Score)
* to describe incidence of bone fractures caused by osteoporosis as well as of other pathological findings of the skeleton after the beginning of the Preotact® treatment
* to describe serum level of calcium and the bone resorption marker desoxypyridinoline (DPD) and N- respectively C-terminal crosslink-telopeptide (CTX and NTX) at the beginning of the Preotact® treatment and at the end of the observational period (only in subgroup of patients, where the physician sees a need to measure these parameters)
* to document all adverse drug reactions after the beginning of the Preotact® treatment
* the analysis of subgroups with different risk for bone fractures caused by osteoporosis at the beginning of the Preotact® treatment
* to assess the manageability and functioning of the Pen system for injection of Preotact® (self administered questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion requires that Preotact® is prescribed in accordance with the SPC and that the stated contraindications are strictly considered.
* Caution should be taken by the treating Physician concerning any precautions, warnings and potential drug interactions stated in the SPC.
* No further inclusion or exclusion parameters are defined. The decision for the individual application of Preotact® will be strictly made by the physicians.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe postmenopausal osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2006-09; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed Deutschland GmbH, Cities in Germany, Germany

REFERENCES:
- [Derived] Moricke R, Rettig K, Bethke TD. Use of recombinant human parathyroid hormone(1-84) in patients with postmenopausal osteoporosis: a prospective, open-label, single-arm, multicentre, observational cohort study of the effects of treatment on quality of life and pain--the PROPOSE study. Clin Drug Investig. 2011;31(2):87-99. doi: 10.2165/11538880-000000000-00000. PMID 21155613